CLINICAL TRIAL: NCT06229639
Title: Assessing the Safety of the Nocturnal Passy Muir Valve and Its Impact on Sleep Quality in an LTACH Setting
Brief Title: Safety of the Nocturnal Passy Muir Valve and Impact on Sleep Quality at an LTACH Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaylord Hospital, Inc (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 201512TAN
Record Dates: First submitted 2023-12-21; First posted 2024-01-29 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Tracheostomy
Keywords: Tracheostomy; Speaking Valve; Sleep Quality; LTACH; Passy-Muir Valve; Respiratory Care
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Tracheostomy Plug (Active Comparator): Patients receive tracheostomy plug during night 2.
  Interventions: Device: Tracheostomy Plug
- Passy-Muir Valve (Experimental): Patients receive Passy-Muir Valve during night 1.
  Interventions: Device: Passy Muir Valve

INTERVENTIONS:
Device: Passy Muir Valve
  Arms: Passy-Muir Valve
Device: Tracheostomy Plug
  Arms: Tracheostomy Plug

SUMMARY:
Limited research has been done to assess the safety of PMV use during sleep. One prospective study completed by Diez-Gross, et al in 2007 looked at 10 male subjects recorded on two consecutive nights, one night with PMV on and one night with PMV off. All recordings took place in a monitored setting. The variables studied included O2 saturation, apnea index, apnea - hypopnea index, and nursing reports. Conclusion was PMV use for one night in seriously ill tracheostomy patients was not associated with respiratory distress or cardiac issues.

DETAILED DESCRIPTION:
Currently, the PMV has only been approved by the FDA for daytime use. As such, it is encouraged to remove speaking valves at night. However, there is minimal evidence indicating that the use of speaking valves during nighttime poses a significant risk. Studies focusing on the safety of the PMV for nocturnal use reported no significant effects on patients' well-being, including no significant oxygen desaturations or major cardiopulmonary events. This was shown in pediatric patients and adult patients admitted to an ICU. While promising, these findings are still limited, and additional evidence is needed to demonstrate the safety of nocturnal PMV use before larger studies can be conducted.

It was anecdotally witnessed that patients frequently sleep during the day with the PMV in place, suffering no recourse to adverse events. The primary objective of this study was to determine if nocturnal PMV use can be considered safe within the long-term acute care hospital setting and its impact on sleep quality

ELIGIBILITY:
Inclusion Criteria:

1. Patient has evidence of respiratory insufficiency requiring a tracheostomy tube without current need for assisted ventilation.
2. Patient will be continuously monitored with telemetry.
3. Patient satisfies criteria for the decannulation protocol and agrees to use the Passy Muir Valve during sleep.
4. Patient is able to follow directions following speech/language/cognitive evaluation or screening completed by the Speech-Language Pathologist and physician assessment.
5. Patient is at least 18 years old.
6. An informed consent is signed by patient or Power of Attorney (POA).
7. Patient is able to tolerate the PMV during the day for a minimum of 6 continuous hours
8. Patient has a maximum size #6 Shiley cuffless tracheostomy tube or equivalent.

Exclusion Criteria:

1. Patient identified at time of admission as requiring invasive long-term assisted ventilation.
2. Patient with documented or suspected upper airway obstruction and/or surgery or permanent tracheostomy tube.
3. Patient is quadriplegic (due to the inability for a quadriplegic patient to manually self-remove the valve in case of emergency).
4. Patient or POA failed to sign consent.
5. Pt has a severe cognitive impairment as determined by a formal cognitive-linguistic evaluation by a licensed Speech Language Pathologist.
6. Patient unable to meet criteria for decannulation protocol or has failed decannulation protocol within last two weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Heart rate | Night 1 at 22:00, 2:00, 6:00 and night 2 at 22:00, 2:00, 6:00
  Measures the number of contractions of the heart per minute (bpm).
Systolic Blood Pressure | Night 1 at 22:00, 2:00, 6:00 and night 2 at 22:00, 2:00, 6:00
  Measures the pressure in your arteries when your heart beats (mmHg).
Diastolic blood pressure | Night 1 at 22:00, 2:00, 6:00 and night 2 at 22:00, 2:00, 6:00
  Measures the pressure in your arteries when your heart rests between beats (mmHg).
Body Temperature | Night 1 at 22:00, 2:00, 6:00 and night 2 at 22:00, 2:00, 6:00
  Measures the normal body temperature of participants (°F).
O2 | Night 1 at 22:00, 2:00, 6:00 and night 2 at 22:00, 2:00, 6:00
  Oxygen saturation measures percentage of oxyhemoglobin in the blood (%).
ETCO2 | Night 1 at 22:00, 2:00, 6:00 and night 2 at 22:00, 2:00, 6:00
  The level of carbon dioxide that is released at the end of an exhaled breath (mm Hg).
Respiratory Rate | Night 1 at 22:00, 2:00, 6:00 and night 2 at 22:00, 2:00, 6:00
  Measures the breathing rate by number of breaths per minute (bpm).

SECONDARY OUTCOMES:
PCO2 | Morning after night 1 and morning after night 2
  The amount of carbon dioxide in the blood in the arterial blood gas measurements (mm Hg).
PO2 | Morning after night 1 and morning after night 2
  The amount of oxygen in the blood by the arterial blood gas measurements (mm Hg).
Bicarbonate | Morning after night 1 and morning after night 2
  The amount of bicarbonate in the blood by the arterial blood gas measurements (mmol/L).
Sleep Quality | Morning after night 1 and morning after night 2
  This is measured by the Richards-Campbell Sleep Questionnaire, which is recorded on a 100 nm visual scale with higher scores indicating better sleep levels than lower scores.
pH | Morning after night 1 and morning after night 2
  The amount of pH in the blood measured by the arterial blood gas measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaylord Hospital, Wallingford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Durbin CG Jr. Tracheostomy: why, when, and how? Respir Care. 2010 Aug;55(8):1056-68. PMID 20667153
- [Background] Lian S, Teng L, Mao Z, Jiang H. Clinical utility and future direction of speaking valve: A review. Front Surg. 2022 Sep 8;9:913147. doi: 10.3389/fsurg.2022.913147. eCollection 2022. PMID 36157432
- [Background] Liney T, Dawson R, Seth R, et al. Anxiety levels amongst patients with tracheostomies. British Journal of Anaesthesia. 2019;123(4):e504-e505. doi:10.1016/j.bja.2019.04.027
- [Background] O'Connor LR, Morris NR, Paratz J. Physiological and clinical outcomes associated with use of one-way speaking valves on tracheostomised patients: A systematic review. Heart Lung. 2019 Jul-Aug;48(4):356-364. doi: 10.1016/j.hrtlng.2018.11.006. Epub 2018 Dec 17. PMID 30573194
- [Background] Passy V, Baydur A, Prentice W, Darnell-Neal R. Passy-Muir tracheostomy speaking valve on ventilator-dependent patients. Laryngoscope. 1993 Jun;103(6):653-8. doi: 10.1288/00005537-199306000-00013. PMID 8502098
- [Background] Winters B, Serpas D, Fullmer N, Hughes K, Kincaid J, Rosario ER, Schnakers C. Sleep Quality Should Be Assessed in Inpatient Rehabilitation Settings: A Preliminary Study. Brain Sci. 2023 Apr 25;13(5):718. doi: 10.3390/brainsci13050718. PMID 37239190
- [Background] DuBose JR, Hadi K. Improving inpatient environments to support patient sleep. Int J Qual Health Care. 2016 Oct;28(5):540-553. doi: 10.1093/intqhc/mzw079. Epub 2016 Aug 10. PMID 27512130
- [Background] Martin JL, Fiorentino L, Jouldjian S, Josephson KR, Alessi CA. Sleep quality in residents of assisted living facilities: effect on quality of life, functional status, and depression. J Am Geriatr Soc. 2010 May;58(5):829-36. doi: 10.1111/j.1532-5415.2010.02815.x. PMID 20722819
- [Background] Shuman AG, Duffy SA, Ronis DL, Garetz SL, McLean SA, Fowler KE, Terrell JE. Predictors of poor sleep quality among head and neck cancer patients. Laryngoscope. 2010 Jun;120(6):1166-72. doi: 10.1002/lary.20924. PMID 20513034
- [Background] 510(k) Premarket Notification. U.S. Food and Drug Administration. Accessed June 23, 2022. https://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfpmn/pmn.cfm?ID=K962714
- [Background] Barraza GY, Fernandez C, Halaby C, Ambrosio S, Simpser EF, Pirzada MB, Islam S. The safety of tracheostomy speaking valve use during sleep in children: a pilot study. Am J Otolaryngol. 2014 Sep-Oct;35(5):636-40. doi: 10.1016/j.amjoto.2014.04.011. Epub 2014 May 4. PMID 24888795
- [Background] Gross RD, Atwood C. R168: Safety of Tracheostomy Speaking Valve Use during Sleep. Otolaryngol Head Neck Surg. 2007;137(2_suppl):P209-P209. doi:10.1016/j.otohns.2007.06.505
- [Background] Richards KC, O'Sullivan PS, Phillips RL. Measurement of sleep in critically ill patients. J Nurs Meas. 2000 Fall-Winter;8(2):131-44. PMID 11227580
- [Background] Silveira AR, Soki MN, Chone CT, Tah Y Ng R, Carvalho EG, Crespo AN. Brazilian tracheotomy speech valve: diaphragm pressure standardization. Braz J Otorhinolaryngol. 2009 Jan-Feb;75(1):107-10. doi: 10.1016/s1808-8694(15)30840-5. PMID 19488569